CLINICAL TRIAL: NCT02596438
Title: Thousand Asian American Study (TAAS)
Brief Title: Thousand Asian American Study
Acronym: TAAS
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 388325
Record Dates: First submitted 2015-10-19; First posted 2015-11-04 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — Hepatitis B Vaccines

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Asian Americans: Foreign born or children of foreign born Asian American from Hepatitis B endemic areas residing in Sacramento, CA.
  Interventions: Other: Hepatitis B

INTERVENTIONS:
Other: Hepatitis B — Hepatitis B Surface Antigen, Hepatitis B Surface Antibody and Hepatitis B Core AB, Total Testing

SUMMARY:
The "Thousand Asian American Study" or "TAAS" aims to test 2,000 foreign-born and children of foreign born Asian Americans residing in Sacramento county residents for HBV and (2) counsel at least 90% of those whose screening results are positive for HBV.

DETAILED DESCRIPTION:
The "Thousand Asian American Study" or "TAAS" aims to better understand the factors associated with testing for hepatitis B viral (HBV) testing among foreign-born Asian and African adult residents of Sacramento county, characteristics of those infected with HBV, and the efficacy of follow-up and linkage to care for those infected with HBV, and develop a research platform for future studies. Thus, what the investigators want to do is 1) test 2000 foreign-born Sacramento county residents for HBV and (2) counsel at least 90% of those whose screening results are positive for HBV. The investigators want to better characterize factors associated with HBV testing and factors that may differentiate those determined to be free of infection, infected with HBV, and those with resulting primary liver cancer.

ELIGIBILITY:
Inclusion Criteria:

* All foreign-born Asians and any foreign-born adults born in CDC-defined high to intermediate endemic areas residing in Sacramento County, California.

Exclusion Criteria:

* Individuals who have been previously serologically tested for Hepatitis B (self-reported).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Asian Americans residing in Sacramento, CA who are 18 years of age and older.
Sampling Method: Non-Probability Sample
Enrollment: 1076 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Number of patients or adult children of patients born in Hepatitis B endemic countries (rate of 2% or higher) getting screened for hepatitis B. | 1 year

SECONDARY OUTCOMES:
Number of patients that are hepatitis B positive that receive counseling regarding their infection. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Moon S Chen Jr., PhD, Principal Investigator — UC Davis Comprehensive Cancer Center
Locations (1):
- University of California, Davis Comprehensive Cancer Center, Sacramento, California, United States

REFERENCES:
- [Derived] Stewart SL, Dang JH, Torok NJ, Chen MS Jr. Patterns and co-occurrence of risk factors for hepatocellular carcinoma in four Asian American communities: a cross-sectional study. BMJ Open. 2019 Jun 28;9(6):e026409. doi: 10.1136/bmjopen-2018-026409. PMID 31256022